CLINICAL TRIAL: NCT04810806
Title: Immediate Versus Delayed Coronary Angiography in Patients With Non-ST-Segment Acute Coronary Syndrome With Acute Decompensated Heart Failure
Brief Title: Timing of Coronary Angiography in NSTE-ACS With ADHF
Acronym: EARLY-HF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Chonnam National University Hospital (Other)
Responsible Party: Principal Investigator, Min Chul Kim, Associate Professor, Chonnam National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNUH-2020-396
Record Dates: First submitted 2021-03-14; First posted 2021-03-23 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure; Acute Coronary Syndrome
Keywords: Heart Failure; Acute Coronary Syndrome; Non-ST-Segment Elevation Acute Coronary Syndrome; Myocardial Infarction; Coronary Disease; Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Heart Failure; Acute Coronary Syndrome; Myocardial Infarction; Coronary Disease; Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate coronary angiography group (Experimental): Immediate coronary angiography group will routinely receive coronary angiography within 2 hours after randomization.
  Interventions: Procedure: Immediate coronary angiography within 2 hours after randomization
- Delayed coronary angiography group (Active Comparator): Delayed coronary angiography group will receive coronary angiography during hospitalization after stabilization of symptoms and signs of heart failure.
  Interventions: Procedure: Delayed coronary angiography after stabilization of heart failure

INTERVENTIONS:
Procedure: Immediate coronary angiography within 2 hours after randomization — After achievement of informed consent in patients with NSTE-ACS complicated by ADHF, patients will be screened and randomized. Patients will be randomized to immediate CAG group or delayed CAG group. Immediate CAG group will receive CAG within 2 hours after randomization. Patients will receive treatment methods according to CAG results: percutaneous coronary intervention (PCI), coronary artery bypass graft (CABG) or medical therapy only by operators' discretion.
  Arms: Immediate coronary angiography group
Procedure: Delayed coronary angiography after stabilization of heart failure — After achievement of informed consent in patients with NSTE-ACS complicated by ADHF, patients will be screened and randomized. Patients will be randomized to immediate CAG group or delayed CAG group. Delayed CAG group will receive CAG after stabilization of ADHF; improvement of symptoms and signs of heart failure. Patients will receive treatment methods according to CAG results: percutaneous coronary intervention (PCI), coronary artery bypass graft (CABG) or medical therapy only by operators' discretion.
  Arms: Delayed coronary angiography group

SUMMARY:
The investigators hypothesized that immediate coronary angiography (CAG) within 2 hours after admission can reduce mortality compared to delayed CAG after stabilization of acute decompensated heart failure (ADHF) in patients with non-ST-segment elevation acute coronary syndrome (NSTE-ACS) complicated by ADHF. Patients with NSTE-ACS complicated by ADHF will be randomized to immediate CAG (coronary angiography < 2 hours after randomization) or delayed CAG after stablization group by 1:1 fashion. This study is a prospective, non-blinded, randomized trial.

DETAILED DESCRIPTION:
Study objective In this study, investigators aim to compare early coronary angiography (CAG < 2 hours after randomization) and delayed CAG after stabilization of acute decompensated heart failure (ADHF) in patients with acute non-ST-elevation acute coronary syndrome (NSTE-ACS) complicated by ADHF. This study is a prospective, non-blinded, randomized trial.

Study background An ADHF is frequently encountered in patients with NSTE-ACS. Although its incidence has been decreased during the decades, it is still high up to 8-12% at initial presentation of NSTE-ACS. Patients with NSTE-ACS complicated by ADHF is also known to be associated with worse in-hospital and long-term clinical outcomes than those without heart failure (HF). Because revascularization could reduce mortality in these patients, it should be done in all patients with NSTE-ACS with ADHF. Current guidelines recommend immediate CAG within 2 hours after admission in patients with NSTE-ACS complicated by ADHF. However, it is difficult to decide the timing of coronary angiography in these high risk patients.

Notably, the most of randomized trials about the timing of coronary angiography in NSTE-ACS excluded these high risk patients, therefore there is lack of evidence for immediate coronary angiography within 2 hours after admission in patients with NSTE-ACS complicated by ADHF.

Investigators will compare immediate CAG within 2 hours after admission and delayed CAG after stabilization of ADHF in patients with NSTE-ACS complicated by ADHF by randomized controlled trial.

Study hypothesis Immediate CAG within 2 hours after admission can reduce mortality compared to delayed CAG after stabilization of ADHF in patients with NSTE-ACS complicated by ADHF.

ELIGIBILITY:
Inclusion Criteria:

1. Age more than 18 years old
2. NSTE-ACS*
3. Pulmonary congestion or edema on chest X-ray

   * The definition of NSTE-ACS

Among patients with typical angina, dyspnea or chest discomfort without definite non-cardiac causes, at least 1 presentations of angina that suggest a NSTE-ACS:

1. Rest angina, which is usually more than 20 minutes in duration
2. New onset angina that markedly limits physical activity
3. Increasing angina that is more frequent, longer in duration, or occurs with less exertion than previous angina

A 12-lead electrocardiogram should have no ST-segment elevation. Cardiac troponin may elevate (non-ST-segment elevation myocardial infarction) or not elevate (unstable angina pectoris).

Exclusion Criteria:

1) Cardiogenic shock* 2) Heart failure of other causes rather than NSTE-ACS 3) Terminal malignancy 4) Life expentancy < 1 year 5) Pregnancy or lactation

* The definition of cardiogenic shock All these criteria should be met

1. Systolic blood pressure < 90 mmHg for 30 minutes, or needing inotropics or vasopressor to maintain systolic blood pressure > or = 90 mmHg
2. Pulmonary congestion on chest X-ray or increased left ventricular filling pressure by cardiac catheterization
3. At least one criteria of organ dysfunction - mental obtundation, clammy ski, ogliuria, renal dysfunction, increased level of blood lactate

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence rate of all-cause death, non-fatal myocardial infarction or recurrent ischemia | Up to 12 months
  Cumulative incidence rate of all-cause death, non-fatal myocardial infarction or recurrent ischemia

SECONDARY OUTCOMES:
Rate of all-cause death, non-fatal myocardial infarction or recurrent ischemia | Up to 12 months
  All-cause death, non-fatal myocardial infarction or recurrent ischemia during initial hospitalization
In-hospital mortality | Up to 12 months
  All-cause mortality during initial hospitalization
In-hospital cardiac mortality | Up to 12 months
  Cardiac mortality during initial hospitalization
Rate of procedural complications during coronary angiography or percutaneous coronary intervention | Up to 12 months
  Rate of procedural complications during coronary angiography or percutaneous coronary intervention during initial hospitalization
Peak level of troponin-I | Up to 12 months
  Peak level of troponin-I during initial hospitalization
Rate of recurrent ischemia | Up to 12 months
  Rate of recurrent ischemia during initial hospitalization
Rate of Non-fatal myocardial infarction | Up to 12 months
  Non-fatal myocardial infarction during initial hospitalization
Rate of stroke | Up to 12 months
  Rate of stroke during initial hospitalization
Usage rate of non-invasive positive pressure ventilation | Up to 12 months
  Usage rate of non-invasive positive pressure ventilation during initial hospitalization
Usage rate of mechanical ventilator | Up to 12 months
  Usage rate of mechanical ventilator during initial hospitalization
Usage rate of renal replacement therapy | Up to 12 months
  Usage rate of renal replacement therapy during initial hospitalization
Usage rate of mechanical circulatory support | Up to 12 months
  Usage rate of mechanical circulatory support during initial hospitalization
Rate of acute kidney injury | Up to 12 months
  Rate of acute kidney injury during initial hospitalization
Rate of stent thrombosis | Up to 12 months
  Rate of stent thrombosis during initial hospitalization
Rate of major bleeding | Up to 12 months
  Rate of major bleeding during initial hospitalization (BARC classificiation 3-5)
Duration of initial hospitalization | Up to 12 months
  Duration of initial hospitalization (days)
Cumulative incidence rate of all-cause death, non-fatal myocardial infarction or recurrent ischemia | Up to 1 month
  Cumulative incidence rate of all-cause death, non-fatal myocardial infarction or recurrent ischemia
Cumulative incidence rate of all-cause death | Up to 1 month
  Cumulative incidence rate of all-cause death
Cumulative incidence rate of cardiac death | Up to 1 month
  Cumulative incidence rate of cardiac death
Cumulative incidence rate of rehospitalization due to heart failure | Up to 1 month
  Cumulative incidence rate of rehospitalization due to heart failure
Cumulative incidence rate of cardiogenic shock | Up to 1 month
  Cumulative incidence rate of cardiogenic shock
Cumulative incidence rate of stroke | Up to 1 month
  Cumulative incidence rate of stroke
Cumulative incidence rate of stent thrombosis | Up to 1 month
  Cumulative incidence rate of stent thrombosis
Cumulative incidence rate of major bleeding (BARC classification 3-5) | Up to 1 month
  Cumulative incidence rate of major bleeding (BARC classification 3-5)
Cumulative incidence rate of recurrent ischemia | Up to 1 month
  Cumulative incidence rate of recurrent ischemia
Cumulative incidence rate of non-fatal myocardial infarction | Up to 1 month
  Cumulative incidence rate of non-fatal myocardial infarction
Cumulative incidence rate of all unplanned revascularization | Up to 1 month
  Cumulative incidence rate of all unplanned revascularization
Cumulative incidence rate of all-cause death | Up to 12 months
  Cumulative incidence rate of all-cause death
Cumulative incidence rate of cardiac death | Up to 12 months
  Cumulative incidence rate of cardiac death
Cumulative incidence rate of rehospitalization due to heart failure | Up to 12 months
  Cumulative incidence rate of rehospitalization due to heart failure
Cumulative incidence rate of cardiogenic shock | Up to 12 months
  Cumulative incidence rate of cardiogenic shock
Cumulative incidence rate of stroke | Up to 12 months
  Cumulative incidence rate of stroke
Cumulative incidence rate of stent thrombosis | Up to 12 months
  Cumulative incidence rate of stent thrombosis
Cumulative incidence rate of major bleeding (BARC classification 3-5) | Up to 12 months
  Cumulative incidence rate of major bleeding (BARC classification 3-5)
Cumulative incidence rate of recurrent ischemia | Up to 12 months
  Cumulative incidence rate of recurrent ischemia
Cumulative incidence rate of non-fatal myocardial infarction | Up to 12 months
  Cumulative incidence rate of non-fatal myocardial infarction
Cumulative incidence rate of all unplanned revascularization | Up to 12 months
  Cumulative incidence rate of all unplanned revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Min Chul Kim, Professor, Principal Investigator — Chonnam National University Hospital
Locations (1):
- Chonnam National University Hospital, Gwangju, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lim Y, Park S, Joo D, Lee YK, Oh S, Lee SH, Ahn JH, Hyun DY, Cho KH, Sim DS, Hong YJ, Kim JH, Ahn Y, Kim MC. Immediate versus delayed coronary angiography in patients with non-ST segment elevation acute coronary syndrome complicated with acute decompensated heart failure: The EARLY-HF randomized clinical trial. Cardiovasc Revasc Med. 2025 Oct 6:S1553-8389(25)00509-3. doi: 10.1016/j.carrev.2025.09.016. Online ahead of print. PMID 41073186